CLINICAL TRIAL: NCT00380939
Title: A Prospective, Randomized, Double-Blind, Multi-Center Study Comparing the Effects of Atorvastatin Versus Pravastatin on the Progression and Quantification of Coronary Atherosclerotic Lesions as Measured by Intravascular Ultrasound (REVERSAL)
Brief Title: This Study Uses Ultrasound to Determine Whether Atorvastatin or Pravastatin Effects the Progression of Coronary Plaque.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0981-400-314
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Coronary Arteriosclerosis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atorvastatin; Pravastatin

INTERVENTIONS:
Drug: Atorvastatin
Drug: Pravastatin

SUMMARY:
This study was designed to assess the effects on coronary artery plaque using aggressive lipid-lowering therapy versus moderate lipid-lowering therapy. A substudy will examine the effect of these treatments on brachial artery vasoactivity.

ELIGIBILITY:
Inclusion Criteria:

* Angiographic evidence of coronary artery disease as defined by a lesion that has at least 20% reduction in luman diameter by visual (angiographic) estimation in any native coronary artery. LDL cholesterol equal to 125mg/dl - 210mg/dl.

Exclusion Criteria:

* Patients who are anticipated to undergo coronary bypass surgery or cardiac transplantation during the course of the study. Known major hematologic, neoplastic, metabolic, gastrointestinal or endocrine dysfunction.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 1999-04; Study Completion 2000-12

PRIMARY OUTCOMES:
The primary efficacy parameter is the percent change in total plaque volume for all slices of anatomically comparable segments of the target coronary artery from baseline to month 18.
The primary efficacy parameter for brachial artery vasoactivity is the nominal change (month 3 - baseline) in the percent arterial diameter change.

SECONDARY OUTCOMES:
The nominal change (month 18 - baseline) in total plaque volume as measured by the sum of plaque areas for all slices of anatomically comparable segments of the target coronary artery.
Changes in brachial artery vasoactivity will be correlated with changes in total cholesterol, LDL-C, triglyceride and apolipoprotein B levels following 3 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- United States (33):
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, BLUE Island, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Shawnee Mission, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Auburn, Maine
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Royal Oak, Michigan
  - Pfizer Investigational Site, Saint Clair, Michigan
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Greensboro, North Carolina
  - Pfizer Investigational Site, Greenville, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Elryia, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Seattle, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0981-400-314&StudyName=This+study+uses+ultrasound+to+determine+whether+atorvastatin+or+pravastatin+effects+the+progression+of+coronary+plaque%2E